CLINICAL TRIAL: NCT05418790
Title: A Pilot Study to Evaluate Alternative Viral Load Tests During Start of Antiretroviral Therapy in Persons Living With HIV: Reliability and Acceptability of Home Test Measures
Brief Title: A Pilot Study to Evaluate Alternative Viral Load Tests During Start of Antiretroviral Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Luis Montaner (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Luis Montaner, Sponsor Investigator, The Wistar Institute
Organization: The Wistar Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: TASSO starting ART
Record Dates: First submitted 2022-06-09; First posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: HIV-1-infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TASSO device (Experimental): During this trial, participants will have approximately 15 TASSO collection dates between in clinic and at home.
  Interventions: Device: TASSO device

INTERVENTIONS:
Device: TASSO device — During this trial, participants will have approximately 15 TASSO collection dates between in clinic and at home.

SUMMARY:
A pilot study of alternative viral load testing with samples collected in the clinic and at home compared to traditional viral load monitoring in participants engaged in HIV care. Approximately 15 participants starting ART, or working to suppress a detectable viral load, will monitor viral loads during regular clinic appointments and in intermediate time-points during their participation in this pilot study.

DETAILED DESCRIPTION:
A pilot study of alternative viral load testing with samples collected in the clinic and at home compared to traditional viral load monitoring in participants engaged in HIV care. Approximately 15 participants starting ART, or working to suppress a detectable viral load, will monitor viral loads during regular clinic appointments and in intermediate time-points during their participation in this pilot study.

There are three planned research viral load evaluations in the trial, which may include but are not limited to the evaluations listed below:

1. CLINICAL CARE VIRAL LOAD - This will take place at the clinic during the regular clinical follow-up to confirm effective viral suppression.. During these visits an HIV viral load sample will be collected using traditional venipuncture methods and analyzed using a qualified commercial test. These plasma values may be used as a comparator with other viral load test results.
2. CLINIC TASSO COLLECTION - Participants will collect one or more Tasso device specimen(s) during in-clinic study visits. The main objective of these measurements is to evaluate HIV viral load monitoring using novel collection approaches with the supervision of trained study staff to minimize user error potential.
3. HOME TASSO COLLECTION - Participants will be provided with Tasso devices to use at home in between regular parent study visits. These devices will be shipped in real-time to Wistar Institute for archiving before HIV viral loads will be measured. The main objective of these measurements is to evaluate the feasibility HIV viral load monitoring using novel collection approaches at home.

ELIGIBILITY:
Inclusion Criteria:

* Persons living with HIV starting an ART regimen or working to suppress a previously detectable viral load ≥ 5,000 copies/mL

Exclusion Criteria:

* Persons living with HIV suppressed on ART regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Reliability and Accuracy | 12 months
  Determine the reliability and accuracy of alternative viral load tests to detect changes in viral load in participants starting ART or working to resuppress a detectable viral load ≥ 5,000 copies/mL at last measurement.
Feasibility of implementing a home-based viral load test | 12 months
  Determine the feasibility of implementing a home-based viral load test in the context of starting ART or working to resuppress a detectable viral load ≥10,0005,000 copies/mL at last measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Montaner, Principal Investigator — The Wistar Institute

IPD SHARING:
Plan to Share IPD: No